CLINICAL TRIAL: NCT03530813
Title: Role of Technology in Improving Asthma Management In School Staff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sydney Children's Hospitals Network (Other)
Responsible Party: Principal Investigator, Stephanie Francis, Paediatric Registrar, Sydney Children's Hospitals Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LNR/15/SCHN/455
Record Dates: First submitted 2018-04-12; First posted 2018-05-21 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Asthma in Children
Keywords: School; Management; Technology; Asthma Education

STUDY DESIGN:
Intervention Model Description: Prospective Randomised Parallel Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-To-Face Group (Active Comparator): Asthma First Aid Management in Schools 3 Hour Face to Face Training Group, selected a training session to attend in their local area.
  Interventions: Other: Face-To-Face Asthma First Aid in Schools Training
- Ebook Group (Experimental): Asthma Management in Schools eBook training group were sent a cloudStor link to download and complete training
  Interventions: Other: Ebook Asthma First Aid in School Training

INTERVENTIONS:
Other: Ebook Asthma First Aid in School Training — Technology assisted, self-directed learning eBook resource
  Arms: Ebook Group
Other: Face-To-Face Asthma First Aid in Schools Training — School Asthma First Aid Management Program 3 Hour Face to Face Training
  Arms: Face-To-Face Group

SUMMARY:
The Asthma First Aid Management for School Staff eBook has been developed for the purpose of providing a multimedia self-directed training resource for school staff. The eBook will be accessible to both primary and secondary school staff; it has the advantage over conventional face to face training in that it can be used for learning when convenient, regardless of geographical location. The eBook has been designed to provide school staff with an alternative training option in contrast to a structured time scheduled face to face asthma first aid management training session. The content of the eBook is based on the information from the current Sydney Children's Hospital, Aiming for Asthma Improvement in Children "School Champion Asthma Management Program" (SCAMP) face to face training course.

This study has been designed to determine the effectiveness of the eBook in meeting the asthma first aid management training needs of school staff, prior to its implementation and uploading to the Apple iBook store where it will be freely available to school staff internationally.

The study will involve school staff being randomized into one of the following two training groups:

Group 1 - a three hour face to face School Champion Asthma Management Program training session (Standard training; control group) Group 2 - completion of the self-directed Asthma First Aid Management for School Staff eBook (Technology assisted learning) The school staff will be required to complete pre and post training validated asthma knowledge questionnaires which will measure improvements in knowledge and confidence. In addition, demographic data will be collected.

The researchers hypothesize that the eBook will provide school staff with an alternative mode of training that will effectively increase school staff asthma management knowledge and confidence. We aim to investigate if this training is superior to the current three hour face to face School Champion Asthma Management Program training.

DETAILED DESCRIPTION:
1. STUDY SITE

   Sydney Children's Hospital High Street Randwick Sydney Australia
2. FUNDING AND RESOURCES

   Existing funding from the Aiming for Asthma Improvement in Children Program (Chronic & Complex Care program, Ministry of Health) general cost centre has been used for the development of resources and to support existing staff FTE's.
3. INTRODUCTION/BACKGROUND INFORMATION

   3.1 INTRODUCTION The Aiming for Asthma Improvement in Children (AAIC) program has been funded by the Ministry of Health as part of the NSW Chronic Disease Program. Its mission is to improve the management of paediatric asthma through provision of standardised resources, education and training, and promotion of best practice strategies, resulting in a specialist coordinated paediatric asthma management service that facilitates continuity of care between hospital and community services.

   AAIC has well established health professional led asthma management training programs for hospital clinicians and community groups which include public and private schools; childcare services; and out of school hours care services. The School Champion Asthma Management Program (SCAMP), implemented in 2010, is one example.

   Based on the work of Professor Richard Henry in the Hunter Region of NSW the SCAMP model adopts a train the trainer approach with a designated school staff member attending a face to face SCAMP cluster training session and taking on the role as School Asthma Champion for their school. With ongoing support from AAIC, the School Asthma Champion facilitates feedback of asthma first aid information to staff within their school as well as facilitating the implementation and maintenance of best practice school asthma management procedures. The designated School Asthma Champion is an important communication link between the school, student, parent, & AAIC. To date, 138 schools have participated in SCAMP with 77 schools having a current SCAMP trained School Asthma Champion.

   Because the train the trainer is resource intensive and presents a barrier to training Schools in remote and rural NSW, we have developed an eBook which will be downloadable from the Apple iBook store. This has the advantage of being more convenient and accessible to any School in NSW (and internationally) if they have an internet connection and an Apple tablet or phone. Prior to its launch we propose to undertake this this study to evaluate its effectiveness.

   3.2 BACKGROUND INFORMATION

   Asthma is a very common disease affecting children in Australia. There are over two million Australians who have been diagnosed with Asthma and 1 in 10 children have been diagnosed with the disease. The New South Wales Child Death Review Team found that 20 children in NSW alone died from asthma between 2004 and 2013 with the number of deaths from asthma in children unexpectedly increasing between 2010 and 2012.

   School teachers are functioning as the carer for children with asthma when they are on school grounds. As children spend on average 30% of their day in school it is clearly vital that these teachers have the necessary knowledge and self-confidence to recognise and manage regarding the symptoms of asthma. This requires both a theoretical understanding of the disease process and a practical understanding of recognising signs of disease and administering first aid treatment.

   It is known that education of both patients and their carers is critical for improving clinical outcomes. We currently have a face-to-face SCAMP training session for educating school teachers about Asthma in place. However, it is resource intensive and does not allow participation of Schools in rural and remote regions. In order to address these issues, we have developed an eBook educational tool for school teachers based on this SCAMP training session and is planned for implementation in 2016. The SCAMP program general feedback has been very positive however we have not formally had the opportunity of evaluating the program in a research setting, hence this proposed study is timely.

   A review of the literature demonstrates that education programs targeting school teachers can be effective in increasing knowledge and awareness about asthma in school children, however formal evaluation of school asthma education programs such as SCAMP, particularly in Australia, is lacking.

   Furthermore, no evaluation has been undertaken using technology assisted learning, such as an electronic book to train school teachers in first aid asthma management which is the aim of this study. There are also no studies directly comparing the efficacy of asthma education between face-to-face education and technology-assisted education.

   If this study demonstrates effectiveness then it is likely to help with uptake from teachers in Schools in Australia and other English speaking countries. It is crucial to undertake the evaluation before publishing the iBook in the Apple store in order to reduce bias during the planned study due to potential access of the control group.
4. STUDY OBJECTIVES 4.1 RESEARCH QUESTION Does technology assisted learning using an iBook increase school staff knowledge and confidence in school asthma first aid management greater than face-to-face training? The hypothesis of the study is that describing asthma first aid knowledge by the SCAMP iBook is superior to standard face to face training.

   4.2 PRIMARY OBJECTIVES

   • To determine if the SCAMP iBook increases school staff asthma management knowledge more than the current face-to-face training.

   4.3 SECONDARY OBJECTIVES

   • To evaluate the usefulness of the SCAMP eBook as a self-directed multi-media teaching resource
5. STUDY DESIGN

   5.1 STUDY TYPE & DESIGN & SCHEDULE

   This is a prospective randomised parallel study, coordinated by SCH AAIC and conducted across NSW schools.

   The target population will be primary and secondary school staff currently employed in a NSW public or private school, who meet the inclusion criteria.

   Participants will be recruited to the study as outlined below and randomised into one of two training groups:

   Group 1 - a 3 hour face to face School Champion Asthma Management Program training session Group 2 - completion of the self-directed SCAMP iBook.

   Randomisation will be done within each school to ensure equal matching of schools demographics in both arms of the study.

   To meet the primary objective of the study, the validated Asthma First Aid Knowledge Questionnaire will be completed prior to and following training.

   To meet the secondary objectives, a 4 item 10 point Likert Scale asthma management self-confidence questionnaire will be completed prior to and following training.

   Surveys will be pre-numbered, consecutively i.e. 1, 2, 3 and randomly distributed to participants, therefore any teacher could get any survey number.

   Surveys will be emailed to teachers allocated to Group 2, and the survey number will initially be recorded against email addresses however, this will be securely destroyed once all surveys are distributed and returned.

   The surveys themselves contain no identifying data.

   All data will only be accessible by the research team, named on this application. Data will be saved on a password-protected hospital drive. No identifiable or re-identifiable data will be published.

   For Group 1 the appropriate forms will be provided before and after the education session. Once completed these forms will be collected and stored as detailed in 11.1, 11.2, & 11.3 of this protocol.

   For Group 2 the Pre Training questionnaires will be sent via email to all participants. These will need to be completed and returned via email within one week of the sent date. We will then send the secure link via email to the iBook along with the Post Training questionnaires. These questionnaires will need to be completed and returned via email within one week of the sent date. Once completed these forms will be collected and stored as detailed below.

   This study will predominantly be conducted at centralised health care facility venues and some NSW school locations.

   5.2 RANDOMISATION

   Once the participating schools with at least 2 willing participants have been identified we will randomize the participating school teachers within each school into either Group 1 or Group 2 using an online randomization tool (HTTPS://www.randomizer.org).

   5.3 STUDY METHODOLOGY

   This study does not involve clinical or laboratory assessment. Data will be collected through self-administered questionnaires, pre and post training. The questionnaires will be collected before and after the face to face training.
6. STUDY POPULATION 6.1 RECRUITMENT PROCEDURE

Study participants will be school staff currently employed in a NSW primary or secondary school, who meet the inclusion criteria as listed elsewhere in the application.

Recruitment will be coordinated as follows:

1. Engagement of primary and secondary school education key stakeholders (DEC, AIS, & CEC) to assist in the promotion of the study to NSW school principals and encourage staff participation
2. AAIC to send follow up invitational email to school principals outlining overview of study, participation involvement and inclusion criteria, and copy of consent form for perusal.
3. On receipt of acceptance by the school principal for school to participate, AAIC to forward recruitment form with options of training dates / times / venues, for staff to select their preferred training date.
4. Upon receipt of the registrations one of the investigators will contact the participant by phone or email in order to determine whether they are appropriate for the study (ie ensure they meet inclusion criteria and do not meet exclusion criteria)
5. The principle investigator will then randomly assign each participant within each school using the on-line random number generator to either Group 1 (Standard training; control group) or Group 2 (Technology assisted learning).
6. Informed consent to participate in study will then be undertaken.

   6.2 CONSENT In addition to receiving HREC approval from SCHN, we will need to receive HREC approval from each of the Educational bodies. Informed written consent that reflect both the education agency Ethics Committee Policy and the SCHN Ethics Committee Policy will be obtained from all participants at the commencement of the study. Participants can withdraw from the study at any time.

   Participants who wish to waive their consent at the commencement of training or withdraw at any time during the study will not be included in the collection or publishing of data but will be able to continue to undertake training in school asthma first aid management via SCAMP face to face cluster training.
7. PARTICIPANT SAFETY AND WITHDRAWAL 7.1 RISK MANAGEMENT AND SAFETY This is a low and negligible risk study. It will involve school staff participating in either face to face asthma management training or self-directed technology assisted asthma management training that they have agreed to undertake for the purpose of professional development. They will be required to complete questionnaires immediately prior to commencing the training and immediately at the completion of the training. We do not anticipate any risks associated with the study as it aims to benefit staff through improved training and support of participants. All care will be taken to deliver ongoing support to participants during and following school asthma first aid management training.

   7.2 HANDLING OF WITHDRAWALS Should at any stage a participant withdraws from the study, the relevant data collected pertaining to the individual will be securely destroyed.

   7.3 REPLACEMENTS Withdrawn participants will be replaced if the number of total participants falls below the target number required for statistical significance.
8. STATISTICAL METHODS

   8.1 SAMPLE SIZE ESTIMATION & JUSTIFICATION

   The hypothesis of the study is that describing asthma first aid knowledge by the SCAMP iBook is superior to standard face to face training.

   The primary outcome measure, asthma first aid knowledge, and will be assessed by the Asthma First Aid Knowledge Questionnaire which has been developed and validated by Dr Bandana Saini and Kate Luckie at the University of Sydney. These validation studies have not yet been published and form part of Kate Luckie's PhD's thesis. In collaboration with the Faculty of Pharmacy, University of Sydney we will be utilising this questionnaire with their kind permission to assess the primary outcome.

   8.2 POWER CALCULATIONS Based on our current data and information from Dr Saini, the sample size is 44 participants required both pre and post intervention in both groups. This calculation is based on the 14-item version of the questionnaire where the pre-intervention score is 11.18± SD 2.5(n=205). Assuming that post face-to-face training there is a 10% improvement (i.e. expecting the final score in group 1 to be 12.68± SD 2.5), and that post iBook there is a further 10% improvement (i.e. expecting the final score in group 2 to be 13.95± SD 2.5), 44 participants in both pre and post intervention are required to demonstrate a significant change with a 80% power and significant set at a 2 sided 5% value.

   Assuming a 15% drop out rate post intervention we aim to recruit 55 participants in each arm.

   8.3 STATISTICAL METHODS TO BE UNDERTAKEN A paired t-test will be utilized to assess pre-post scores and Likert scales.
9. DATA SECURITY & HANDLING

9.1 DETAILS OF WHERE RECORDS WILL BE KEPT & HOW LONG WILL THEY BE STORED Data collected as a hard copy will be stored in a locked cupboard, in an office in the Respiratory Department of Sydney Children's Hospital Randwick. Data entered electronically will be saved in the AAIC folder on the SCHN Network F drive, which is password protected. All data collected will be stored for a minimum of 7 years with disposal by secure shredding or electronic erasure consistent with the SCHN correct disposal of secure information policy.

9.2 CONFIDENTIALITY AND SECURITY Information provided by participants and their associated schools will only be accessible to members of the research team. Published data will be de-identified to maintain confidentiality. Written notification of confidentiality and security will be documented on the consent form of which recruited school staff will have a copy.

ELIGIBILITY:
Inclusion Criteria:

* Currently employed as a school staff member in NSW public,private,catholic school
* Available to attend a 3 hour training session if randomly assigned to group
* Access to ipad, mac pc or iphone with iphone application installed
* Literate in English language

Exclusion Criteria

- previously participated in SCAMP

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2016-08-12 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2016-12-14 (Actual)

PRIMARY OUTCOMES:
Change in Asthma First Aid Knowledge Questionnaire Knowledge (AFAKQ) Questionnaire | Group1 Pre-questionnaire completed onsite at training, prior to commencement & post completed immediately following 3hour training. Group 2 PreQuestionniare emailed 1 wk prior to ebook link being sent & post to be completed within 3 wks of receiving link
  AFAKQ is a 14 item validated questionnare developed and validated by the University Of Sydney, Australia. Faculty Of Pharmacy

SECONDARY OUTCOMES:
Change in Asthma Management Self-Confidence Questionnaire | Group1 Pre-questionnaire completed onsite at training, prior to commencement & post completed immediately following 3hr training. Group 2 PreQuestionniare emailed 1 wk prior to ebook link being sent & post to be completed within 3 wks of receiving link
  4 item, 10 point Likert Scale- Self reported skill confidence in emergency asthma mangement . Value no.0 represented as being not confident at all with a scale moving towards the Value no. 10 representing very confident

CONTACTS AND LOCATIONS:
Overall Officials: Professor Adam Jaffe, BSc(Hons) MD, Principal Investigator — University Of New South Wales. Australia
Locations (1):
- Sydney Childrens Hospital Network, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henry RL, Hazell J, Halliday JA. Two hour seminar improves knowledge about childhood asthma in school staff. J Paediatr Child Health. 1994 Oct;30(5):403-5. doi: 10.1111/j.1440-1754.1994.tb00688.x. PMID 7833074
- [Background] Hazell J, Henry RL, Francis JL, Halliday JA. Teacher initiated improvement of asthma policy in schools. J Paediatr Child Health. 1995 Dec;31(6):519-22. doi: 10.1111/j.1440-1754.1995.tb00875.x. PMID 8924303
- [Background] Henry RL, Gibson PG, Vimpani GV, Francis JL, Hazell J. Randomized controlled trial of a teacher-led asthma education program. Pediatr Pulmonol. 2004 Dec;38(6):434-42. doi: 10.1002/ppul.20095. PMID 15690558
- [Background] Fitzgerald DA, Gillis J. Asthma deaths in children in New South Wales 2004-2013: Could we have done more? J Paediatr Child Health. 2015 Nov;51(11):1127-33. doi: 10.1111/jpc.12947. Epub 2015 Jul 1. PMID 26135337
- [Background] Wesseldine LJ, McCarthy P, Silverman M. Structured discharge procedure for children admitted to hospital with acute asthma: a randomised controlled trial of nursing practice. Arch Dis Child. 1999 Feb;80(2):110-4. doi: 10.1136/adc.80.2.110. PMID 10325723
- [Background] Wolf FM, Guevara JP, Grum CM, Clark NM, Cates CJ. Educational interventions for asthma in children. Cochrane Database Syst Rev. 2003;2002(1):CD000326. doi: 10.1002/14651858.CD000326. PMID 12535395
- [Background] Kawafha MM, Tawalbeh LI. The effect of asthma education program on knowledge of school teachers: a randomized controlled trial. West J Nurs Res. 2015 Apr;37(4):425-40. doi: 10.1177/0193945914528070. Epub 2014 Mar 29. PMID 24682383
- [Background] Soo YY, Saini B, Moles RJ. Can asthma education improve the treatment of acute asthma exacerbation in young children? J Paediatr Child Health. 2013 May;49(5):353-60. doi: 10.1111/j.1440-1754.2012.02551.x. Epub 2012 Sep 12. PMID 22970747
- [Background] Shah S, Gibson PG, Wachinger S. Recognition and crisis management of asthma in schools. J Paediatr Child Health. 1994 Aug;30(4):312-5. doi: 10.1111/j.1440-1754.1994.tb00652.x. PMID 7946541
- [Background] McWhirter J, McCann D, Coleman H, Calvert M, Warner J. Can schools promote the health of children with asthma? Health Educ Res. 2008 Dec;23(6):917-30. doi: 10.1093/her/cym081. Epub 2008 Mar 5. PMID 18325911